CLINICAL TRIAL: NCT01128777
Title: Mental Health Intervention for Teens Coping With Parental Military Deployment
Brief Title: Teens Coping With Parental Military Deployment
Acronym: Helping Hand
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to difficuly recruiting participants
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH082164 (NIH); R34MH082164 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Emotional Distress; Behavior Problems
Keywords: depression; anxiety; family conflict; behavior problems
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive behavioral group therapy (Experimental): Cognitive behavioral group therapy for adolescents and a parallel group for parents
  Interventions: Behavioral: Cognitive Behavioral Group Therapy
- Nondirective supportive group therapy (Active Comparator): Nondirective supportive group therapy for adolescents and a parallel group for parents
  Interventions: Behavioral: Nondirective supportive group therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy — The CBT group therapy protocol will teach adolescents coping, cognitive restructuring, and affect regulation skills to remediate skills deficits that underlie depression, anxiety, and behavior problems associated with the deployment cycle. Parents will also learn stress management and parenting skills in their own group therapy sessions that occur as the same time as the adolescent group.
  Arms: Cognitive behavioral group therapy
Behavioral: Nondirective supportive group therapy — Patient initiated discussions form the basis for the intervention for both the adolescent group and the parent group
  Arms: Nondirective supportive group therapy

SUMMARY:
The total number of military personnel is over 3.5 million and approximately 43% have children. The deployment cycle can be associated with depression, anxiety, and behavior problems in children as well as psychological distress in the military spouse. Further, the health of family members can affect the physical and psychological functioning of the military service member during the deployment and re-integration periods. While research and federal funding has been dedicated toward developing treatments for the returning service member, intervention protocols for mental health problems in the children of military families have not been tested. In collaboration with the Family Readiness Program of the Rhode Island National Guard & Reserves, the purpose of this proposal is to develop a cognitive behavioral treatment protocol for adolescents experiencing depression, anxiety, and/or behavior problems associated with the deployment and re-integration phases of the military deployment cycle. This protocol will be created by modifying an NIH funded cognitive behavioral protocol for the treatment of adolescent mental health problems with initial demonstrated efficacy (PI, C. Esposito-Smythers). There are three primary aims in this project: 1) develop the manualized intervention protocol for adolescents experiencing mental health problems associated with the deployment cycle; 2) refine and pilot the intervention protocol with 12 families; and 3) test the intervention in a randomized pilot trial. To accomplish these aims, a two step sequence of treatment development is proposed. Stage Ia includes initial manual development, focus groups, therapist training, and an open pilot trial. Stage Ib includes a randomized pilot trial. Seventy-two adolescents and their caretakers will be enrolled through the Rhode Island Family Readiness program and randomly assigned to the experimental intervention or non-directive supportive therapy for their outpatient care. The experimental intervention includes 12 adolescent group sessions which address depression, anxiety, and behavior problems associated with the deployment cycle and 12 parent group sessions that address stress management and parenting skills. The non-directive supportive therapy condition includes 12 adolescent and 12 parent group sessions which involve patient initiated discussions focused on issues surrounding military deployment and re-integration. Outcome will be assessed at post-treatment and 3 month follow-up. The long term objective of this research is to yield an effective outpatient intervention for teens of military service members experiencing mental health problems associated with the deployment and re-integration phases of the deployment cycle.

ELIGIBILITY:
Inclusion Criteria:

Adolescents must: 1) be 13-17 years old; 2) be English speaking; 3) provide adolescent assent; 4) have parental consent and a parent/legal guardian available to participate in the intervention protocol; 5) have a parent who is deployed or returned from a deployment within the last year; and 6) report current sub-clinical or clinical levels of depression, anxiety, or oppositional behavior. In order to meet the symptom criterion, adolescents must receive a T score of ≥ 65 on the affective problems, anxiety problems, and/or oppositional defiant problems on the Youth Self-Report or the Child Behavior Checklist.

Exclusion Criteria:

Adolescents who : 1) are developmentally delayed such that the intervention materials will not be appropriate; 2) are actively suicidal or psychotic at intake; 3) are receiving pharmacotherapy or psychotherapy in the community for depression, anxiety, or disruptive behavior which are the primary targets of this intervention; or 4) meet current criteria for a DSM-IV diagnosis of bipolar disorder, conduct disorder, substance dependence, or obsessive-compulsive disorder.

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Depressed mood | baseline, posttreatment, 3 month follow-up

SECONDARY OUTCOMES:
Behavior problems | baseline, posttreatment, 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Brown Univerity, Providence, Rhode Island, United States